CLINICAL TRIAL: NCT00218920
Title: Effective Training in Overweight and Obesity
Brief Title: Effective Training in Overweight and Obese People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2005.542
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Overweight
Keywords: aerobic capacity; endothelial function; exercise
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- strength training (Experimental): Over a 12-week period, 13 subjects performed three programmed exercise sessions per week; two supervised by the study investigators in the research laboratory and one performed at home or in a gym, according to instructions.
  Interventions: Behavioral: Strength training
- continuous moderate-intensity aerobic training (Experimental): Over a 12-week period, 13 subjects performed three programmed exercise sessions per week; two supervised by the study investigators in the research laboratory and one performed at home or in a gym, according to instructions.
  Interventions: Behavioral: continuous moderate-intensity aerobic training
- high-intensity interval aerobic training (Experimental): Over a 12-week period, 14 subjects performed three programmed exercise sessions per week; two supervised by the study investigators in the research laboratory and one performed at home or in a gym, according to instructions.
  Interventions: Behavioral: high-intensity interval aerobic training

INTERVENTIONS:
Behavioral: Strength training — a strength training regime of 4 series with 5 repetitions each, at approximately 90% of 1 repetition maximum (RM), in a leg press apparatus to develop maximal strength mainly from neural adaptation with minimal weight gain due to muscular hypertrophy.
  Arms: strength training
Behavioral: continuous moderate-intensity aerobic training — The moderate-intensity group walked continuously for 47 min at 60-70% of maximum heart rate (HRmax) to ensure that the training protocols were isocaloric.
  Arms: continuous moderate-intensity aerobic training
Behavioral: high-intensity interval aerobic training — High-intensity training consisted of a 10 min warm-up period at 50-60% of HRmax [maximal HR (heart rate)], followed by 4×4-min intervals at 85-95% of HRmax with 3 min active breaks in between the intervals, consisting of walking or jogging at 50-60% of HRmax. The exercise session was terminated by a 5 min cool-down period.
  Arms: high-intensity interval aerobic training

SUMMARY:
The aim is to come to a consensus about how to prescribe exercise training that actually helps overweight and obese people. Thus, the present study determines the effects of several types of exercise training to define the one with the largest effect with the least effort.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) over 30

Exclusion Criteria:

* Not able to walk on a treadmill
* Participating in an other study
* Serious cardiovascular diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 weeks
Aerobic capacity | 12 weeks
Endothelial function | 12 weeks

SECONDARY OUTCOMES:
Molecular markers in fat and skeletal muscle biopsies for the effects of exercise training | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Schjerve IE, Tyldum GA, Tjonna AE, Stolen T, Loennechen JP, Hansen HE, Haram PM, Heinrich G, Bye A, Najjar SM, Smith GL, Slordahl SA, Kemi OJ, Wisloff U. Both aerobic endurance and strength training programmes improve cardiovascular health in obese adults. Clin Sci (Lond). 2008 Nov;115(9):283-93. doi: 10.1042/CS20070332. PMID 18338980